CLINICAL TRIAL: NCT04551469
Title: A Randomized Clinical Trial to Measure Efficacy of Music on Cardiac Surgery
Brief Title: A Randomized Clinical Trial to Measure Efficacy of Music on Cardiac Surgery Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Diane L. Carroll, nurse researcher, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MusicCS
Record Dates: First submitted 2020-09-03; First posted 2020-09-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Surgery
Keywords: music; cardiac surgery; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): 30 minutes of listening to music
  Interventions: Behavioral: music
- Standard of Care (No Intervention): actual sounds of the intensive care unit environment

INTERVENTIONS:
Behavioral: music — Music intervention for 30 minutes
  Arms: Treatment Arm

SUMMARY:
Cardiac surgery involves both physical and psychological stress for patients from time of decision to the recovery period. The physical aspects and the impact on the psychological experience makes the post-operative period a difficult time for patients. Patients often experience emotional distress, uncertainty, and fear. A non-pharmacological intervention of music may affect the patient's perception of early recovery with little to no side effects.

Current research has demonstrated efficacy in psychological and physical responses. there is limited data on the endocrinologic (cortisol) and immunologic biomarkers Immunoglobulin A to a music intervention. Therefore, the purpose of this study is to measure both psychological/physical response and biomarkers pre and post a 30-minute music intervention compared to standard of care experience A randomized, placebo-controlled, pre-post clinical trial will be initiated to demonstrate the effect that music has on the primary outcome of serum cortisol and secondary outcomes of anxiety, pain, blood pressure, heart rate, respirations, and Immunoglobulin A in adult patients after cardiac surgery.

DETAILED DESCRIPTION:
One hundred-twelve subjects will be enrolled, 56 subjects in the treatment and 56 subjects in the standard of care group. It was estimated this sample size would be needed to detect a medium effects size of .30 with an alpha set at a level of .05.

Patients, who agree to participate, will be randomly allocated to one of two groups, treatment and standard of care group using a computer-generated randomization scheme.

On post-operative day one, two or three, a 30-minute music period will be used through personal headphones and a MP3 device. Music will be a selection that is symphonic music that has no dramatic changes. The standard of care group will listen to environmental sounds in the Cardiac Surgical Intensive Care Unit.

Psychological, and physical responses as well as biomarkers will be collected pre and then 30 minutes after the start of the intervention period in both groups. The psychological response will be assessed by the Spielberger State Anxiety Scale to measure state anxiety and a visual analogue scale for measurement of pain. Physical responses will be collected that includes Blood pressure in mmHg, heart rate in beats per minute and respirations in beats per minute. The biomarkers collected will be serum cortisol measured in micrograms per deciliter and Immunoglobulin in milligrams per deciliter.

Descriptive statistics will be used to describe the sample and the outcomes measure will be compared using a student t-test.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the Cardiac Surgical Intensive Care Unit or the Cardiac Surgical Step Down Unit after undergoing heart valve replacement/repair and/or coronary artery bypass surgery, or aortic repair over the age of 18 years, hemodynamically stable, extubated and able to hear music.

Exclusion Criteria:

* Patients that are deaf, hemodynamically unstable, intubated, and on infectious disease precautions after surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Cortisol | Change in serum cortisol before and 30 minutes after start of intervention period
  micrograms per deciliter

SECONDARY OUTCOMES:
Anxiety | Change in state anxiety before and 30 minutes after start of intervention period
  Spielberger State Anxiety Scale (STAI) -2 0 to 80 with higher score more Anxiety.
Perceived Pain Level | Change in pain level before and 30 minutes after start of intervention period
  Visual Analogue Pain Scale- 0 to 10 with 0 = no pain to 10=worst pain.
Blood Pressure | Change in blood pressure before and 30 minutes after start of intervention period
  mm Hg
Heart Rate | Change in heart rate before and 30 minutes after start of intervention period
  beats per minute
Respirations | Change in respirations before and 30 minutes after start of intervention period
  breaths per minute
Serum Immunoglobulin A | Change in serum immunoglobulin A before and 30 minutes after start of intervention period
  mg per deciliter

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wahbeh H, Haywood A, Kaufman K, Zwickey H. Mind-Body Medicine and Immune System Outcomes: A Systematic Review. Open Complement Med J. 2009;1:25-34. doi: 10.2174/1876391X00901010025. PMID 23227136
- [Background] Finn S, Fancourt D. The biological impact of listening to music in clinical and nonclinical settings: A systematic review. Prog Brain Res. 2018;237:173-200. doi: 10.1016/bs.pbr.2018.03.007. Epub 2018 May 1. PMID 29779734
- [Background] Nilsson U. The effect of music intervention in stress response to cardiac surgery in a randomized clinical trial. Heart Lung. 2009 May-Jun;38(3):201-7. doi: 10.1016/j.hrtlng.2008.07.008. Epub 2008 Oct 5. PMID 19486788
- [Background] Chlan LL, Weinert CR, Heiderscheit A, Tracy MF, Skaar DJ, Guttormson JL, Savik K. Effects of patient-directed music intervention on anxiety and sedative exposure in critically ill patients receiving mechanical ventilatory support: a randomized clinical trial. JAMA. 2013 Jun 12;309(22):2335-44. doi: 10.1001/jama.2013.5670. PMID 23689789
- [Background] Liu Y, Petrini MA. Effects of music therapy on pain, anxiety, and vital signs in patients after thoracic surgery. Complement Ther Med. 2015 Oct;23(5):714-8. doi: 10.1016/j.ctim.2015.08.002. Epub 2015 Aug 4. PMID 26365452
- [Background] Heidari S, Babaii A, Abbasinia M, Shamali M, Abbasi M, Rezaei M. The Effect of Music on Anxiety and Cardiovascular Indices in Patients Undergoing Coronary Artery Bypass Graft: A Randomized Controlled Trial. Nurs Midwifery Stud. 2015 Dec;4(4):e31157. doi: 10.17795/nmsjournal31157. Epub 2015 Dec 1. PMID 26835471